CLINICAL TRIAL: NCT04149574
Title: A Phase 3, Randomized, Double-blind Trial of Nivolumab in Combination With Intravesical BCG Versus Standard of Care BCG Alone in Participants With High-risk Non-muscle Invasive Bladder Cancer That Is Persistent or Recurrent After Treatment With BCG
Brief Title: A Study Comparing the Efficacy and Safety of Nivolumab in Combination With Bacillus Calmette-Guerin (BCG) Versus BCG Alone in Participants With High-Risk Non-Muscle Invasive Bladder Cancer (HR NMIBC)
Acronym: CheckMate 7G8
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient enrollment, inability to meet protocol objectives, and slow accrual.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-7G8
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: nivolumab + Bacillus Calmette-Guérin (BCG) (Experimental)
  Interventions: Drug: nivolumab; Biological: Bacillus Calmette-Guérin (BCG)
- Arm B: placebo +BCG (Placebo Comparator)
  Interventions: Other: Placebo; Biological: Bacillus Calmette-Guérin (BCG)

INTERVENTIONS:
Drug: nivolumab — Specified Dose on Specified Days
  Arms: Arm A: nivolumab + Bacillus Calmette-Guérin (BCG)
Other: Placebo — Specified Dose on Specified Days
  Arms: Arm B: placebo +BCG
Biological: Bacillus Calmette-Guérin (BCG) — Specified Dose on Specified Days

SUMMARY:
A study comparing nivolumab and bacterial drugs given to help the body's immune system in the bladder versus bacterial drugs alone in high risk bladder cancer participants.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or recurrent disease ≤ 24 months of last BCG dose, but not classified as BCG unresponsive
* Histologically confirmed persistent or recurrent high-risk non-muscle-invasive urothelial carcinoma (UC)
* Treated with at least 1 adequate course of induction BCG therapy (at least 5 out of 6 doses)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2

Exclusion Criteria:

* Previous or concurrent muscle invasive, locally advanced, or disseminated/metastatic UC
* UC in the upper genitourinary tract (kidneys, renal collecting systems, ureters) within 24 months of enrollment
* UC and/or CIS in the prostatic urethra within 12 months of enrollment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (63):
- United States (2):
  - The University Of Chicago, Chicago, Illinois
  - Local Institution - 0084, The Bronx, New York
- Argentina (7):
  - Local Institution - 0009, Caba, Buenos Aires
  - Local Institution - 0088, Capital Federal, Buenos Aires
  - Local Institution - 0016, Ciudad Autonoma Beunos Aires, Buenos Aires
  - Local Institution - 0081, Mar del Plata, Buenos Aires
  - Local Institution - 0008, Viedma, Río Negro Province
  - Local Institution - 0080, Buenos Aires
  - Local Institution - 0107, Córdoba
- Australia (3):
  - Local Institution - 0002, Sydney, New South Wales
  - Local Institution - 0001, Woolloongabba, Queensland
  - Local Institution - 0114, Bowral
- Austria (4):
  - Local Institution - 0097, Linz
  - Local Institution - 0104, Salzburger
  - Local Institution - 0099, Vienna
  - Local Institution - 0098, Wels
- Brazil (4):
  - Local Institution - 0050, Uberlândia, Minas Gerais
  - Local Institution - 0048, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0047, Itajaí, Santa Catarina
  - Local Institution - 0049, Rio de Janeiro
- Canada (4):
  - Local Institution - 0017, Toronto, Ontario
  - Local Institution - 0038, Montreal, Quebec
  - Local Institution - 0037, Montreal, Quebec
  - Local Institution - 0012, Rimouski, Quebec
- Chile (3):
  - Local Institution - 0011, La Serena, Coquimbo Region
  - Local Institution - 0072, Viña del Mar, Región de Valparaíso
  - Local Institution - 0010, Recoleta, Santiago Metropolitan
- France (8):
  - Local Institution - 0042, Angers
  - Local Institution - 0106, Dijon
  - Local Institution - 0045, Lille
  - Local Institution - 0108, Marseille
  - Local Institution - 0111, Paris
  - Local Institution - 0103, Paris
  - Local Institution - 0041, Strasbourg
  - Local Institution - 0040, Villejuif
- Germany (4):
  - Local Institution - 0105, Cologne
  - Local Institution - 0094, Herne
  - Local Institution - 0093, Jena
  - Local Institution - 0095, Trier
- Greece (2):
  - Local Institution - 0031, Haidari
  - Local Institution - 0032, Thessaloniki
- Israel (3):
  - Local Institution - 0075, Tel Aviv, Tel Aviv
  - Local Institution - 0073, Jerusalem
  - Local Institution - 0074, Ramat Gan
- Italy (6):
  - Local Institution - 0067, Torino, TO
  - Local Institution - 0062, Milan
  - Local Institution - 0063, Modena
  - Local Institution - 0064, Napoli
  - Local Institution - 0065, Reggio Emilia
  - Local Institution - 0066, Roma
- Netherlands (2):
  - Local Institution - 0054, Arnhem
  - Local Institution, Rotterdam
- Russia (2):
  - Local Institution - 0051, Moscow
  - Local Institution - 0052, Saint Petersburg
- Spain (7):
  - Local Institution - 0096, Pamplona, Navarre
  - Local Institution - 0061, Badajoz
  - Local Institution - 0060, Badalona-barcelona
  - Local Institution - 0055, Madrid
  - Local Institution - 0059, Sabadell
  - Local Institution - 0057, Santander
  - Local Institution - 0058, Valencia
- Sweden (2):
  - Local Institution - 0087, Norrköping
  - Local Institution - 0083, Umeå

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study terminated shortly after phase 1 (safety period), phase 2 efficacy period did not initiate.
Groups:
- Arm A: Nivolumab 480 mg intravenous (IV) every 4 weeks (Q4W) for up to 24 months (104 weeks) and intravesical BCG (induction) weekly for 6 weeks followed by maintenance intravesical BCG weekly for 3 weeks at 3, 6, 12, 18, 24, 30, and 36 months
- Arm B: Nivolumab-placebo IV Q4W for up to 24 months (104 weeks) and intravesical BCG (induction) weekly for 6 weeks followed by maintenance intravesical BCG weekly for 3 weeks at 3, 6, 12, 18, 24, 30, and 36 months
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (9.8) | 73.0 (15.3) | 65.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Event Free Survival
Description: The time between the date of randomization and the date of first documented event or death due to any cause, whichever occurs first. Events include recurrence of disease (TaHG, T1, or CIS) and progression of disease.
  Data Not Collected (DNC)
Time Frame: Approximately 44 Months and 1 Week
Population: Study terminated. Data Not Collected. Study was terminated due to slow enrollment. Decision was made to terminate study before entering phase 2 (efficacy portion).
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Part 2: Worsening-Free Survival
Description: The time from randomization to progression to muscle-invasive disease (ie, T2), cystectomy, systemic chemotherapy, radiotherapy, or death from any cause.
  Data Not Collected (DNC)
Time Frame: Approximately 44 months and 1 week
Population: as for outcome 1
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Part 2: Overall Survival
Description: The time between the date of randomization and the date of death due to any cause. For participants still alive, OS is censored at the last date the participant is known to be alive.
  Data Not Collected (DNC)
Time Frame: Approximately 44 months and 1 week
Population: as for outcome 1
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Part 2: Complete Response Rate at 13 Weeks
Description: CRR is defined as the proportion of participants with CIS (+/- TaHG/T1) per PRC at randomization who are disease free at the first disease assessment (Week 13)
  Data Not Collected (DNC)
Time Frame: 13 Weeks
Population: as for outcome 1
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Part 2: Duration of Response
Description: the time between the date of the first CR to the date of first documented recurrence, progression, or death due to any cause.
  Data Not Collected (DNC)
Time Frame: Approximately 44 months and 1 week
Population: as for outcome 1
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: All-causality Adverse Events Leading to Discontinuation
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
  Grading will be based on NCI CTCAE version 5.0 criteria.
Time Frame: 24.6 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 8 | 4
Participants
  Any Grade | 1 | 3
  Grade 3-4 | 0 | 0
  Grade 5 | 0 | 0

7. Secondary Outcome: All-causality Adverse Events
Description: as for outcome 6
Time Frame: 24.6 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 8 | 4
Participants
  Grade 1 | 1 | 2
  Grade 2 | 4 | 1
  Grade 3 | 1 | 1

8. Secondary Outcome: Drug-related Adverse Events
Description: as for outcome 6
Time Frame: 24.6 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 8 | 4
Participants
  Grade 1 | 1 | 1
  Grade 2 | 4 | 1
  Grade 3 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 100 days): Approximately 44 months and 1 week All-Cause mortality (From randomization to end of study): Approximately 44 months and 1 week
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/4
Other Adverse Events (participants affected / at risk) | 5/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=8) | Arm B (N=4)
Cystitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=8) | Arm B (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyschezia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Cortisol decreased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 3 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Immune-mediated cystitis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT04149574/Prot_SAP_000.pdf